CLINICAL TRIAL: NCT07357844
Title: Pediatric Optimal Tuberculosis Treatment Evaluation and Reassessment
Acronym: POTTER
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 25-5044
Record Dates: First submitted 2025-07-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis Disease
Keywords: Tuberculosis; Children
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2014-2024: Historical group, retrospectively described in 2025
- 2025-2026: Post-structuring of the pediatric infectious diseases' activity group, retrospectively described end of 2026

SUMMARY:
The treatment of tuberculosis disease in children benefits from clear and up-to-date recommendations from the World Health organization. The research issues supported by the WHO mainly concern tuberculosis treatment implementation in areas of high incidence and low economic level. Pediatric cohorts in countries with high economic levels are rare, making it impossible to quantify and describe deviations from optimal recommendations. The French recommendations are mainly focused on screening cases of tuberculosis, without specific guidelines for care organization and recent practice evaluation.

The retrospective study of patients followed by the pediatric infectious disease team of the Hospices Civils de Lyon (HCL) would allow to quantify treatment successes and failures, and to describe these failures in a French pediatric tertiary care center. This retrospective analysis is part of an evolution of the pediatric infectious diseases' activity of HCL in 2024: structuring of the service with a full-time practitioner, establishment of multi-professional care with the involvement of psychologists and clinical pharmacists. This retrospective study will help to understand the causes of failure in French tertiary pediatric centers and to describe the expected benefits of a structured and multi-professional care to improve the treatment of pediatric tuberculosis diseases in France.

ELIGIBILITY:
Inclusion Criteria :

- Patients under 18 years old, with tuberculosis disease confirmed from patient's clinical file

Exclusion Criteria :

* Tuberculosis disease ruled out from patient's clinical file
* Parental opposition or patient opposition (if over 18 years old)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0-18 years treated and followed-up in Hospices Civils de Lyon from 2014 to 2026 by the pediatric infectious diseases team for tuberculosis disease.
  Hospices Civils de Lyon is the sole pediatric tertiary care center and pediatric infectious diseases ward in the county.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tuberculosis treatment outcome | 2014-2024
  Tuberculosis treatment outcome, per World Health organization definitions: failed, cured, completed, died, lost to follow-up, not evaluated, success

SECONDARY OUTCOMES:
Secondary outcomes | 2024-2026
  Compliance with anti-tuberculosis treatment
Secondary outcomes: | 2024-2026
  Compliance with follow-up consultations
Secondary outcomes | 2024-2026
  Adapted anti-tuberculosis treatment dosage
Secondary outcomes | 2024-2026
  Adverse effects attributed to anti-tuberculosis treatment
Secondary outcomes | 2024-2026
  Microbiological failure
Secondary outcomes | 2024-2026
  Extension of treatment
Secondary outcomes | 2024-2026
  Modification of treatment regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, Rhônes, France